CLINICAL TRIAL: NCT06956781
Title: Optimizing Behavioral Health Services Following Pediatric Trauma Exposure
Brief Title: Multiphase Optimization Strategy (MOST) for Treating Pediatric Post-traumatic Stress Disorder (PTSD)
Acronym: MOST for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Chad Shenk, Professor of Psychology, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00010448
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: PTSD; Trauma; Pediatric ALL
Keywords: PTSD; Trauma; Pediatric; Multiphase Optimization Strategy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: 2^4 Full Factorial Randomized Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Independent and masked raters of treatment fidelity; Independent and masked raters of processes of change during active treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Treatment Condition 1 (Experimental): Participants receive emotion regulation, exposure, cognitive processing, and bi-lateral stimulation
  Interventions: Behavioral: Emotion Regulation; Behavioral: Exposure; Behavioral: Cognitive Processing; Behavioral: Bi-lateral Stimulation
- Treatment Condition 2 (Experimental): Participants receive emotion regulation, exposure, cognitive processing, and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Exposure; Behavioral: Cognitive Processing; Behavioral: Psychological Placebo
- Treatment Condition 3 (Experimental): Participants receive emotion regulation, exposure, bi-lateral stimulation, and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Exposure; Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 4 (Experimental): Participants receive emotion regulation, exposure, and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Exposure; Behavioral: Psychological Placebo
- Treatment Condition 5 (Experimental): Participants receive emotion regulation, cognitive processing, bi-lateral stimulation, and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Cognitive Processing; Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 6 (Experimental): Participants receive emotion regulation, cognitive processing, and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Cognitive Processing; Behavioral: Psychological Placebo
- Treatment Condition 7 (Experimental): Participants receive emotion regulation, bi-lateral stimulation, and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 8 (Experimental): Participants receive emotion regulation and psychological placebo
  Interventions: Behavioral: Emotion Regulation; Behavioral: Psychological Placebo
- Treatment Condition 9 (Experimental): Participants receive exposure, cognitive processing, bi-lateral stimulation, and psychological placebo
  Interventions: Behavioral: Exposure; Behavioral: Cognitive Processing; Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 10 (Experimental): Participants receive exposure, cognitive processing, and psychological placebo
  Interventions: Behavioral: Exposure; Behavioral: Cognitive Processing; Behavioral: Psychological Placebo
- Treatment Condition 11 (Experimental): Participants receive exposure, bi-lateral stimulation, and psychological placebo
  Interventions: Behavioral: Exposure; Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 12 (Experimental): Participants receive exposure and psychological placebo
  Interventions: Behavioral: Exposure; Behavioral: Psychological Placebo
- Treatment Condition 13 (Experimental): Participants receive cognitive processing, bi-lateral stimulation, and psychological placebo
  Interventions: Behavioral: Cognitive Processing; Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 14 (Experimental): Participants receive cognitive processing and psychological placebo
  Interventions: Behavioral: Cognitive Processing; Behavioral: Psychological Placebo
- Treatment Condition 15 (Experimental): Participants receive bi-lateral stimulation and psychological placebo
  Interventions: Behavioral: Bi-lateral Stimulation; Behavioral: Psychological Placebo
- Treatment Condition 16 (Experimental): Participants receive psychological placebo
  Interventions: Behavioral: Psychological Placebo

INTERVENTIONS:
Behavioral: Emotion Regulation — Participants learn to reduce acute subjective distress, stabilize negative mood, promote positive mood, and alter physiological responses to trauma
  Arms: Treatment Condition 1; Treatment Condition 2; Treatment Condition 3; Treatment Condition 4; Treatment Condition 5; Treatment Condition 6; Treatment Condition 7; Treatment Condition 8
Behavioral: Exposure — Participants engage in written exercises to reduce avoidance of trauma reminders and reinforce approach behaviors consistent with personal goals
  Arms: Treatment Condition 1; Treatment Condition 10; Treatment Condition 11; Treatment Condition 12; Treatment Condition 2; Treatment Condition 3; Treatment Condition 4; Treatment Condition 9
Behavioral: Cognitive Processing — Participants learn ways to identify, challenge, and overcome the influence of cognitive distortions resulting from trauma exposure
  Arms: Treatment Condition 1; Treatment Condition 10; Treatment Condition 13; Treatment Condition 14; Treatment Condition 2; Treatment Condition 5; Treatment Condition 6; Treatment Condition 9
Behavioral: Bi-lateral Stimulation — Participants engage in horizontal eye movements while recalling a traumatic memory and describing their affective and physiological state
  Arms: Treatment Condition 1; Treatment Condition 11; Treatment Condition 13; Treatment Condition 15; Treatment Condition 3; Treatment Condition 5; Treatment Condition 7; Treatment Condition 9
Behavioral: Psychological Placebo — Participants receive non-directive support therapy, where they will guide the treatment session but not be required to discuss prior trauma exposure
  Arms: Treatment Condition 10; Treatment Condition 11; Treatment Condition 12; Treatment Condition 13; Treatment Condition 14; Treatment Condition 15; Treatment Condition 16; Treatment Condition 2; Treatment Condition 3; Treatment Condition 4; Treatment Condition 5; Treatment Condition 6; Treatment Condition 7; Treatment Condition 8; Treatment Condition 9

SUMMARY:
The goal of this clinical trial is to test the extent to which different treatment components work to improve pediatric post-traumatic stress disorder (PTSD). It will also provide evidence for how these components work. The main research questions are:

What are the effects of different components used to treat PTSD? What do these components change to produce benefits in PTSD?

Researchers will:

Compare components to a psychological placebo to estimate their effects and measure how they work

Examine how components work alone and in conjunction with other components

Participants will:

Receive different combinations of components and placebo

Attend weekly treatment sessions

Provide information to evaluate changes in PTSD

ELIGIBILITY:
Inclusion Criteria:

A child between the ages of 8-17 exposed to at least one DSM-defined trauma

Child assent for participation

The participation of a caregiver with custodial rights to provide parental permission

Willing to participate in treatment delivery and respond to surveys

Meet PTSD diagnostic criteria that is the result of exposure to at least one of the identified traumas

Ability to read and understand English

Willingness to be randomized to an experimental condition

Placement in a stable caregiving environment for two months without an impending transition

Children currently taking psychotropic medications must have taken the medicine without dose adjustment for two months prior to study entry.

Caregiver or child with a smartphone capable of downloading a freely available software application.

Exclusion Criteria:

Psychiatric concerns requiring a higher level of care (e.g. suicidal ideation with intent; current psychotic disorder)

An intelligence quotient (IQ) < 70

Currently receiving a behavioral health intervention for concerns related to PTSD or pediatric trauma

A participating caregiver who is a perpetrator of any identified trauma (e.g. sexual abuse)

MRI contraindicators (e.g. presence of metal in the body)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Mean Change in PTSD Symptoms - Clinician Administered PTSD Scale for DSM-5 - Child/Adolescent Version (CAPS-CA) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CAPS-CA is a clinician-administered diagnostic interview measuring the severity of PTSD symptoms in the past month. The interview assesses 20 PTSD symptoms according to DSM-5 diagnostic criteria with each symptom rated on a severity scale ranging from 0 to 4. Ratings for each individual symptom are summed with higher scores indicating greater severities of PTSD symptoms (total scores range from 0-80).
Mean Change in PTSD Symptoms - Child PTSD Symptom Scale for DSM-5 (CPSS) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CPSS is a child-report survey measuring the severity of PTSD symptoms in the past month. Survey items assess 20 PTSD symptoms according to DSM-5 diagnostic criteria with severity ratings for each item ranging from 0-4. Ratings for each individual symptom are summed with higher scores indicating greater severities of PTSD symptoms (total scores range from 0-80).
Mean Change in PTSD Symptoms - Child and Adolescent Trauma Screen (CATS-2) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CATS-2 is a caregiver-reported survey measuring the frequency of pediatric PTSD symptoms in the past four weeks. Survey items assess 20 PTSD symptoms according to DSM-5 and ICD-11 diagnostic criteria with frequency ratings for each item ranging from 0-3. Ratings for each individual item are summed with higher scores indicating greater frequencies of PTSD symptoms (total scores range from 0-60).

SECONDARY OUTCOMES:
Change in the Number of Participants with a PTSD Diagnosis - The Clinician Administered PTSD Scale for DSM-5 - Child / Adolescent Version (CAPS-CA) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CAPS-CA is a clinician-administered interview establishing the presence of a PTSD diagnosis according to DSM-5 diagnostic criteria. The presence of a PTSD diagnosis (yes/no) will be established before and after receiving treatment. Change in PTSD diagnostic status will be used to indicate treatment response.
Change in PTSD Symptom Trajectories - Child PTSD Symptom Scale for DSM-5 (CPSS) | Baseline (pre-treatment), Weeks 1-18 (active treatment), Week 19 (post-treatment)
  The CPSS is a child-report survey measuring the severity of PTSD symptoms that will be modified to assess these symptoms in the time since the last treatment session. Survey items assess 20 PTSD symptoms according to DSM-5 diagnostic criteria with severity ratings for each item ranging from 0-4. Ratings for each individual symptom are summed with higher scores indicating greater severities of PTSD symptoms (total scores range from 0-80).
Change in PTSD Symptom Trajectories - Child and Adolescent Trauma Screen (CATS-2) | Baseline (pre-treatment), Weeks 1-18 (active treatment), Week 19 (post-treatment)
  The CATS-2 is a caregiver-reported survey measuring the frequency of pediatric PTSD symptoms that will be modified to assess these symptoms in the time since the last treatment session. Survey items assess 20 PTSD symptoms according to DSM-5 and ICD-11 diagnostic criteria with frequency ratings for each item ranging from 0-3. Ratings for each individual item are summed with higher scores indicating greater frequencies of PTSD symptoms (total scores range from 0-60).
Mean Change in Mood Disorder Symptoms - Children's Depression Inventory-2 (CDI-2) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CDI-2 is a child-report survey assessing the severity of twenty-eight mood disorder symptoms in the past two weeks. Responses are rated on a scale from 0-2 and summed. Higher scores indicate greater severities of mood disorder symptoms (total raw scores range from 0-56). Raw scores can be converted to T-scores.
Mean Change in Anxiety Disorder Symptoms - Screen for Child Anxiety Related Disorders (SCARED) | Baseline (pre-treatment, Week 19 (post-treatment)
  The SCARED is a child-report survey assessing symptoms of five pediatric anxiety disorders (panic/somatic, generalized anxiety, separation anxiety, social phobia, and school phobia) in the past three months. Responses assess the presence of 41 anxiety symptoms on a scale ranging from 0-2. Item responses are summed with higher scores indicating more severe anxiety symptoms (total scores range from 0-82).
Mean Change in Disruptive Behavior Disorder Symptoms - Child Behavior Checklist (CBCL) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CBCL is a caregiver-report survey measuring the frequency of child behavior problems in the past six months, including disruptive behavior disorder symptoms. There are 112 items rated on a scale of 0-2 with individual item ratings summed to indicate greater symptom frequency (total scores range from 0-238). Raw scores can be converted to T-scores. The externalizing disorders broadband scale and the DSM-oriented scales will be used to measure disruptive behavior disorder symptoms.
Change in PTSD, Mood, Anxiety, and Disruptive Behavior Disorder Symptom Trajectories - Ecological Momentary Assessment (EMA) | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  A 29-item, once-daily EMA will be administered to children via smartphone application for a period of two-weeks at pre-treatment, mid-treatment, and post-treatment. Items assess the presence and duration of PTSD, mood, anxiety, and disruptive behavior disorder symptoms on a scale from 0-100. Higher scores indicate a longer duration of symptoms experienced for the day the survey is completed.
Changes in Trajectories of C-Reactive Protein (CRP) | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  The Tasso+ device will be used to obtain whole blood samples. Tasso+ is an FDA 510(k)-approved, sterile, disposable blood lancing device approved for use by laypeople (e.g. caregiver, research staff). A sterile lancet punctures the skin with the press of a button that simultaneously creates a slight vacuum to help capillary blood flow into a compatible tube under gravity. Depending on blood yield, CRP will be assayed.
Changes in Trajectories of Interleukin-6 (IL-6) | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  The Tasso+ device will be used to obtain whole blood samples. Tasso+ is an FDA 510(k)-approved, sterile, disposable blood lancing device approved for use by laypeople (e.g. caregiver, research staff). A sterile lancet punctures the skin with the press of a button that simultaneously creates a slight vacuum to help capillary blood flow into a compatible tube under gravity. Depending on blood yield, IL-6 will be assayed.
Changes in Trajectories of Tumor Necrosis Factor-Alpha | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  The Tasso+ device will be used to obtain whole blood samples. Tasso+ is an FDA 510(k)-approved, sterile, disposable blood lancing device approved for use by laypeople (e.g. caregiver, research staff). A sterile lancet punctures the skin with the press of a button that simultaneously creates a slight vacuum to help capillary blood flow into a compatible tube under gravity. Depending on blood yield, tumor necrosis factor-alpha will be assayed.
Brain Aging - Magnetic Resonance Imaging (MRI) | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  MRIs will be performed to measure changes in brain aging, the difference between a participant's chronological age and biological age estimated through several established neural markers. Positive brain aging scores indicate faster brain aging. Negative brain aging scores indicate slower brain aging.
Change in Neural Structure - Magnetic Resonance Imaging (MRI) | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  MRIs will be performed to measure changes in neural structures (e.g. hippocampal and amygdala volume) involved in memory retrieval as well as threat and fear processing associated with PTSD and treatment of PTSD.
Change in Network Connectivity - Magnetic Resonance Imaging (MRI) | Baseline (pre-treatment), A randomly selected two-week period during active treatment (Weeks 5-18), Week 19 (post-treatment)
  MRIs will be performed to measure changes in network connectivity (e.g. default mode network) related to working memory performance, autobiographical recall, and fear processing.
Mean Change in Experiential Avoidance - Avoidance and Fusion Questionnaire for Youth (AFQ-Y) | Baseline (pre-treatment), Week 19 (post-treatment)
  The AFQ-Y is a 17-item child report survey assessing experiential avoidance in the presence of aversive private stimuli. Items are anchored on a 0-4 scale with responses summed to indicate greater levels of avoidance (total scores range from 0-68).
Mean Change in Trauma-Related Cognitions - Child Post-Traumatic Cognitions Inventory (CPTCI) | Baseline (pre-treatment), Week 19 (post-treatment)
  The CPTCI is a 25-item measure assessing the presence of different cognitions that may occur following exposure to pediatric trauma. Each item is ranked on a 1-4 scale with individual responses summed to indicate a greater number of trauma-related cognitions (total scores range from 25-100).
Mean Change in Emotion Transitions - Affect Transition Task | Baseline (pre-treatment), Week 19 (post-treatment)
  Subjects rate the likelihood that a person would transition between two hypothetical affective states. In each trial, subjects are presented with two states connected by an arrow (e.g. happy - angry) and are informed that the state to the left of the arrow is the person's current state and the state on the right side of the arrow is a state the person might experience next. The states included are: hate, love, happy, hurt, mad, sad, scared, and tired. Subjects then rate the likelihood of that person making that transition on a continuous scale from 0-100% with higher scores indicating a greater likelihood of that transition. For a second set of tasks, subjects rate the similarity between each pair of states using a scale from 0-100% with higher ratings indicating greater similarity. Variation in the likelihood ratings for each paired states are examined across participants.
Mean Change Subclinical Psychosis - Prodromal Questionnaire Brief Child Version Screener (PQ-BC) | Baseline (pre-treatment), Week 19 (post-treatment)
  The PQ-BC is a 21-item child-report survey assessing subclinical psychotic symptoms, including unusual beliefs and perceptual distortions in the past month. Each item assesses the presence of a subclinical psychotic symptom in a yes/no response format. A distress score, which weights the endorsed item by the level of distress experienced by that item on a scale of 0-6, is obtained for each of the 21 items. Total scores range from 0-126 with higher scores indicating greater distress.
Mean Change Transdiagnostic Psychiatric Symptoms - The Kiddie Schedule for Affective Disorders and Schizophrenia - Cross Cutting Symptoms (K-SADS-CC) | Baseline (pre-treatment), Week 19 (post-treatment)
  The K-SADS-CC is a 21-item child-report survey assessing psychiatric symptoms common across different psychiatric disorders. Each item assesses the severity of a psychiatric symptom during the past two weeks on a scale of 0-4. Total scores range from 0-84 with higher scores indicating a greater severity of psychiatric symptoms.
Mean Change Transdiagnostic Psychiatric Symptoms - The Kiddie Schedule for Affective Disorders and Schizophrenia - Cross Cutting Symptoms (K-SADS-CC) | Baseline (pre-treatment), Week 19 (post-treatment)
  The NIDA mASSIST is a 15-item child-report survey assessing the use of substances. Each item assesses the frequency of use for a specified substance during the past two weeks on a scale of 0-4. Change in the use of individual substances can be examined over time. A polysubstance use severity score can also be generated by summing the frequencies of all individual items. Total scores for the polysubstance use severity score range from 0-84 with higher scores indicating a greater severity of substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Shenk, PhD, Principal Investigator — University of Rochester
Locations (1):
- The Mt. Hope Family Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and analytic code will be shared on open science outlets
Supporting Information: Analytic Code
Time Frame: De-identified data and statistical code will be shared following closure of the trial and after primary hypotheses have been tested and results published
Access Criteria: Freely available to scientists via open science outlets